CLINICAL TRIAL: NCT02536911
Title: An Open-label Pharmacokinetic and Tolerability Study of Eliglustat Tartrate Given as a Single Dose in Subjects With Mild and Moderate Hepatic Impairment, and in Matched Subjects With Normal Hepatic Function
Brief Title: A Study of the Effects of Hepatic Impairment on the Pharmacokinetics and Tolerability of Eliglustat Tartrate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP13777; U1111-1170-3678 (Other: UTN)
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GZ385660 (healthy subjects) (Experimental): Single dose of eliglustat tartrate will be given under fed conditions
  Interventions: Drug: eliglustat
- GZ385660 (subjects with mild hepatic impairment) (Experimental): Single dose of eliglustat tartrate will be given under fed conditions
  Interventions: Drug: eliglustat
- GZ385660 (subjects with moderate hepatic impairment) (Experimental): Single dose of eliglustat tartrate will be given under fed conditions
  Interventions: Drug: eliglustat

INTERVENTIONS:
Drug: eliglustat — Pharmaceutical form: capsule
  Route of administration: oral
  Other Names: GZ385660

SUMMARY:
Primary Objective:

To study the effect of mild and moderate hepatic impairment on the pharmacokinetics (PK) of eliglustat.

Secondary Objective:

To assess the tolerability of eliglustat tartrate given as a single dose in subjects with mild and moderate hepatic impairment in comparison with matched subjects with normal hepatic function.

DETAILED DESCRIPTION:
The total study duration from screening period is approximately 31 days.

ELIGIBILITY:
Inclusion criteria :

For subjects with hepatic impairment:

* Male or female subjects, between 18 and 79 years of age, inclusive.
* Body weight between 50.0 and 125.0 kg, inclusive if male, and between 40.0 and 110.0 kg, inclusive if female, body mass index (BMI) between 18.0 and 37 kg/m^2, inclusive.
* Stable chronic liver disease assessed by medical history, physical examination, laboratory values.
* For moderate hepatic impairment cohort: Child-Pugh total score ranging from 7 to 9, inclusive.
* For mild hepatic impairment cohort: Child-Pugh total score ranging from 5 to 6, inclusive.

For matched subjects:

* Male or female subjects, between 18 and 79 years of age, inclusive.
* Body weight within 15% of the body weight of the subjects with hepatic impairment and BMI between 18.0 and 37 kg/m^2, inclusive.
* Matched by cytochrome P450 (CYP) 2D6 predicted phenotype based on genotype.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).

Exclusion criteria:

For subjects with hepatic impairment:

* Uncontrolled clinically relevant cardiovascular, pulmonary, gastrointestinal, metabolic, hematological, neurological, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Hepatocarcinoma.
* Acute hepatitis.
* Hepatic encephalopathy grade 2, 3, and 4.
* Presence or history of drug hypersensitivity, or allergic disease, including active seasonal rhinitis, diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day) within 2 years before inclusion.
* If female, pregnancy (defined as positive beta-human chorionic gonadotropin [β -HCG] blood test), breastfeeding.
* P-gp inhibitors and/or inducers, CYP2D6 and/or CYP3A inhibitors and/or inducers.
* Positive result on any of the following tests: anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).
* Pre-existing cardiac disease (current congestive heart failure, recent acute myocardial infarction, bradycardia, heart block, ventricular arrhythmia), long QT syndrome, or use of Class IA (eg, quinidine, procainamide) and Class III (eg, amiodarone, sotalol) anti-arrhythmic medications.
* Any subject with CYP2D6 indeterminate or ultra-rapid metabolizer (URM) phenotype.

For matched subjects:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* If female, pregnancy (defined as positive β-HCG blood test), breastfeeding.
* For subjects 50 years of age and younger: any medication (including St John's Wort) within 14 days before inclusion, or within 5 times the elimination half-life or pharmacodynamic half-life of that medication, whichever the longest, with the exception of hormonal contraception or menopausal hormone replacement therapy, any vaccination within the last 28 days, and any biologics (antibody or its derivatives) given within 4 months before inclusion.
* For subjects older than 50 years of age: any significant change in chronic treatment medication within 14 days before inclusion.
* P-gp inhibitors and/or inducers, CYP2D6 and/or CYP3A inhibitors and/or inducers.
* Positive result on any of the following tests: hepatitis B surface antigen (HBs Ag), anti-hepatitis C virus (anti-HCV) antibodies, anti-HIV1 and anti-HIV2 Ab.
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day) within 2 years before inclusion.
* Pre-existing cardiac disease (current congestive heart failure, recent acute myocardial infarction, bradycardia, heart block, ventricular arrhythmia), long QT syndrome, or use of Class IA (eg, quinidine, procainamide) and Class III (eg, amiodarone, sotalol) anti-arrhythmic medications.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Assessment of PK parameter: Maximum plasma concentration observed (Cmax) | 3 days
Assessment of PK parameter: Area under the plasma concentration (AUC) | 3 days

SECONDARY OUTCOMES:
Assessment of PK parameter: Area under the plasma concentration versus time curve (AUClast) | 3 days
Assessment of PK parameter: Apparent total body clearance (CL/F) | 3 days
Assessment of PK parameter: Apparent volume of distribution during the terminal phase (Vz/F) | 3 days
Assessment of PK parameter: Predicted accumulation ratio (Rac,pred) | 3 days
Assessment of PK parameter: Terminal half-life (t1/2z) | 3 days
Change from baseline in ECG parameter | Baseline, Up to 10 days
Number of adverse events | Up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- United States (2):
  - Investigational Site Number 840002, Miami, Florida
  - Investigational Site Number 840001, Knoxville, Tennessee